CLINICAL TRIAL: NCT02428192
Title: A Phase 2 Study of Nivolumab and Ipilimumab in Advanced Leiomyosarcoma of the Uterus
Brief Title: Nivolumab Alone or in Combination With Ipilimumab in Treating Patients With Advanced Uterine Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02403; NCI-2014-02403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); DFCI- 15-707; 9672 (Other: Dana-Farber - Harvard Cancer Center LAO); 9672 (Other: CTEP); UM1CA186709 (NIH)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Leiomyosarcoma; Unresectable Leiomyosarcoma; Uterine Corpus Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (nivolumab - closed to accrual on 21-Oct-2015) (Experimental): Patients receive nivolumab IV over approximately 60 minutes once every 2 weeks for up to 46 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Nivolumab
- Cohort B (nivolumab and Ipilimumab) (Experimental): Patients receive nivolumab IV over approximately 60 minutes followed by a saline flush and ipilimumab IV over 90 minutes. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Cohort B (nivolumab and Ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Cohort A (nivolumab - closed to accrual on 21-Oct-2015)

SUMMARY:
This phase II trial studies how well nivolumab alone or in combination with ipilimumab works in treating patients with uterine cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment. Monoclonal antibodies, such as nivolumab and ipilimumab, may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of patients with advanced leiomyosarcoma of the uterus (ULMS) treated with nivolumab.

II. To evaluate the objective response rate per RECIST 1.1 of patients with advanced ULMS treated with nivolumab in combination with ipilimumab.

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of nivolumab in patients with advanced ULMS. II. To evaluate the toxicity of nivolumab in combination with ipilimumab in patients with advanced ULMS.

III. To evaluate the progression-free survival of ULMS treated with nivolumab. IV. To evaluate the progression-free survival of ULMS treated with nivolumab in combination with ipilimumab.

V. To explore the relationship between PDL1, PD1 in infiltrating lymphocytes and PD2 status in archival tumor, and pre/post treatment biopsies in a minimum of 10 patients.

TERTIARY OBJECTIVES:

I. To explore the relationship between general immune response and specific markers of immunomodulation and response to nivolumab.

II. To explore the relationship between tumor inflammatory gene signature and response to nivolumab in archival material.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

Cohort A (closed to accrual on 21-Oct-2015): Patients receive nivolumab intravenously (IV) over approximately 60 minutes once every 2 weeks for up to 46 doses in the absence of disease progression or unacceptable toxicity.

Cohort B: Patients receive nivolumab IV over approximately 60 minutes followed by a saline flush and ipilimumab IV over 90 minutes. Treatment repeats every 21 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced leiomyosarcoma of the uterus (ULMS); advanced ULMS is defined as metastatic ULMS or unresectable primary ULMS
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have received at least one prior line of chemotherapy, for ULMS (either in the adjuvant or metastatic setting)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of greater than 9 months
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN/ =< 5 x ULN for subjects with liver metastases
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* Patients with a requirement for steroid treatment or other immunosuppressive treatment: patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 31 weeks after the last dose of investigational drug; women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab; women must not be breastfeeding; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) do not require contraception

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
  * WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; these durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days
  * Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* For enrollment in the first stage of Cohort B, patients must have accessible pre-treatment and post-treatment (4-6 weeks) tumor for biopsy

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (AEs) due to agents administered more than 3 weeks earlier; patients who have had prior pelvic radiation may be at increased risk for bowel perforation, and therefore may not have residual inflammatory disease of the bowel or residual bowel toxicity based on baseline imaging and clinical assessment; palliative (limited-field) radiation therapy is permitted, if all of the following criteria are met:

  * Repeat imaging demonstrates no new sites of bone metastases
  * The lesion being considered for palliative radiation is not a target lesion
  * Bowel toxicity is not expected from the target field due to increased risk of perforation
* Patients who are receiving any other investigational agents
* Patients are excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-ligand 2 (L2), anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Active brain metastasis or leptomeningeal disease; patients with known brain metastases are allowed if metastases have been treated and there is no magnetic resonance imaging (MRI) evidence of progression for at least 12 weeks after treatment is complete and within 28 days prior to the first dose of nivolumab administration; there must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study drug administration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with nivolumab
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) or if they have a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, are excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, fistula and abdominal carcinomatosis should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2021-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015) | Cohort B (Nivolumab and Ipilimumab)
Started | 12 | 8
Completed | 0 | 7
Not Completed | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015) | Cohort B (Nivolumab and Ipilimumab) | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Continuous [Median (Full Range); unit: years] | 54 [29 to 73] | 61 [53 to 76] | 54 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 8 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 8 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Among Patients With Advanced Leiomyosarcoma of the Uterus (ULMS) Treated With Nivolumab (Cohort A)
Description: For the primary endpoint of overall response with a null hypothesis of 5% and an alternative hypothesis of 20%, 37 patients are needed in a two-stage design with 12 patients in the first stage and 25 patients in the second stage. At the first stage analysis, overall response, at least 1 response out of 12 patients will need to be observed to continue through the second stage. At the second stage, at least 4 responses out of 37 patients will need to be observed to accept the treatment. The overall power for overall response rate is 90%. The overall type I error, the chance of incorrectly rejecting the null hypothesis is 9%. The probability of stopping at the first stage under the null hypothesis is 54%. The operating characteristics of this design are calculated using the exact binomial distribution.
Time Frame: Up to 100 days
Population: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015)
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Objective Response Per RECIST 1.1 Among Patients With Advanced ULMS Treated With Nivolumab and Ipilimumab (Cohort B)
Description: For the primary endpoint of overall response with a null hypothesis of 5% and an alternative hypothesis of 30%, 25 patients are needed in a two-stage design with 8 patients in the first stage and 17 patients in the second stage. At the first stage analysis, overall response, at least 1 response out of 8 patients will need to be observed to continue through the second stage. At the second stage, at least 3 responses out of 25 patients will need to be observed to accept the treatment. The overall power for overall response rate is 94%. The overall type I error, the chance of incorrectly rejecting the null hypothesis is 9%. The probability of stopping at the first stage under the null hypothesis is 66%. The operating characteristics of this design are calculated using the exact binomial distribution.
Time Frame: Up to 100 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Nivolumab and Ipilimumab)
Number analyzed (Participants) | 8
Participants | 0

3. Secondary Outcome: Incidence of Toxicity, Graded Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Version 5.0 Beginning April 1, 2018) (Cohort A)
Description: Among the first phase of 12 patients, there is at least 58% probability of observing one or more rare (7% true probability) events, and 83% probability of observing toxicities that have a true occurrence of at least 15%. Among the total cohort of 37 patients, there is at least 85% probability of observing one or more rare (5% true probability) events, and 95% probability of observing toxicities that have a true occurrence of at least 8%. With 37 treated patients, the maximum width of a 90% two-sided exact binomial confidence interval for any estimated adverse event proportion will be no wider than +/- 14%.
Time Frame: Up to 4 cycles
Population: Please see the adverse events module for detailed list of adverse events. Percentage of participants who experienced an adverse event.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015)
Number analyzed (Participants) | 12
Participants | 12

4. Secondary Outcome: Incidence of Toxicity, Graded Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Version 5.0 Beginning April 1, 2018) (Cohort B)
Description: Among the first phase of 8 patients, there is at least 57% probability of observing one or more rare (10% true probability) events, and 73% probability of observing one or more toxicities that have a true occurrence rate as low as 15%. Among the total cohort of 25 patients, there is at least 84% probability of observing one or more rare (7% true probability) events, and 93% probability of observing toxicities that have a true occurrence of at least 10%. With 25 treated patients, the maximum width of a 90% two-sided exact binomial confidence interval for any estimated adverse event proportion will be no wider than +/- 18%.
Time Frame: Up to 4 cycles
Population: Please refer to adverse event module for detailed list of adverse events. Percentage of participants who experienced adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort B (Nivolumab and Ipilimumab)
Number analyzed (Participants) | 8
Participants | 8

5. Secondary Outcome: Rate of Progression-free Survival (Cohort A)
Description: A null hypothesis of 20% and an alternative hypothesis of 40% at 12 weeks will be investigated. Patients lost to follow-up or deaths within 12 weeks will be counted as failures. The overall power for overall progression-free rate at 12 weeks is 87%, using the exact binomial distribution. The operating characteristics of this design are calculated using a one-sided exact test with 10% type I error.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed at 12 weeks
Population: Progression is defined as using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015)
Number analyzed (Participants) | 12
months | 1.8 [0.8 to NA] — The upper limit for the confidence interval on median PFS is unknown because the upper confidence limit for the PFS curve never reached 0.50 hence no upper limit for the median PFS exists.

6. Secondary Outcome: Rate of Progression-free Survival (Cohort B)
Description: A null hypothesis of 18% and an alternative hypothesis of 40% at 6 months will be investigated. Patients lost to follow-up or deaths within 6 months will be counted as failures. The overall power for overall progression-free rate at 6 months is 85%, using the exact binomial distribution. The operating characteristics of this design are calculated using a one-sided exact test with 10% type I error.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed at 6 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort B (Nivolumab and Ipilimumab)
Number analyzed (Participants) | 8
months | 2.0 [0.9 to 2.1]

7. Secondary Outcome: PDL1 Status
Description: The relationship between PDL1 status and response to nivolumab will be explored. A Fisher's exact test will be used to assess the relationship between each biomarker and response to treatment. The power to detect the relationship of interest increases as the prevalence of the biomarker increases.
Time Frame: Up to 100 days
Population: to few responders to analyze biomarker data
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015) | Cohort B (Nivolumab and Ipilimumab)
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: PD2 Status in Archival Tumor
Description: The relationship between PD2 status in archival tumor and response to nivolumab will be explored. A Fisher's exact test will be used to assess the relationship between each biomarker and response to treatment. The power to detect the relationship of interest increases as the prevalence of the biomarker increases.
  Analysis is pending.
Time Frame: Baseline
Reporting Status: Not Posted

9. Other Pre Specified Outcome: PD1 in Infiltrating Lymphocytes
Description: The relationship between PD1 in infiltrating lymphocytes and response to nivolumab will be explored. A Fisher's exact test will be used to assess the relationship between each biomarker and response to treatment. The power to detect the relationship of interest increases as the prevalence of the biomarker increases.
  Analysis is pending.
Time Frame: Up to 100 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 cyles
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events grade 3 or higher per CTCAEv4. Other AEs were defined as anticipated and unanticipated events (not included in the serious adverse event table) that exceed a frequency threshold of 5%. These are grouped by organ system, with number and frequency of such events in each arm/group of the clinical study.
Arm/Group | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015) | Cohort B (Nivolumab and Ipilimumab)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 4/12 | 3/8
Other Adverse Events (participants affected / at risk) | 12/12 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015) (N=12) | Cohort B (Nivolumab and Ipilimumab) (N=8)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Colic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Surgical Procedures (debulking/palliative surgery) (General disorders) | 1 (1) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (Nivolumab - Closed to Accrual on 21-Oct-2015) (N=12) | Cohort B (Nivolumab and Ipilimumab) (N=8)
Akathisia (Nervous system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Chills (General disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 9 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 2 | 0
Edema Limbs (General disorders) | 1 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 8 | 2
Fever (General disorders) | 1 | 1
Flu like Symptoms (General disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 2
Heat Intolerance (Endocrine disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Weight Loss (Investigations) | 3 | 1
White Blood Cell Decreased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Lipase increased (Investigations) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Serum amylase increased (Investigations) | 1 | 1
Stomach pain (Gastrointestinal disorders) | 0 | 1
Abdominal Distention (Gastrointestinal disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 3
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0
Eye disorders - Other, specify - Eye Redness (Eye disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal & urinary disorders - Other - Dysuria (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Resp, thoracic & mediast - Other - Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Resp, thoracic & mediast - Other - Sinus Pressure (Skin and subcutaneous tissue disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Skin & subcutaneous tissue -Other - Skin Sensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Surgical and medical - Other - Debulking/Palliative Surgery (Surgical and medical procedures) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Eye Pain (Eye disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Small Intestine Obstruction (Gastrointestinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Vaginal Dryness (Reproductive system and breast disorders) | 0 | 1
Vaginal Infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02428192/Prot_SAP_000.pdf